CLINICAL TRIAL: NCT05535907
Title: BOLT Lithotripsy RESTORE BTK Trial for PAD (RESTORE BTK)
Brief Title: BOLT Lithotripsy RESTORE BTK Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bolt Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-001700
Record Dates: First submitted 2022-09-03; First posted 2022-09-10 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Disease
Keywords: PAD
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, non- randomized, multi-center study for treatment of stenotic lesions with the Bolt Intravascular Lithotripsy system
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Intravascular lithotripsy (Experimental)
  Interventions: Device: Intravascular Lithotripsy

INTERVENTIONS:
Device: Intravascular Lithotripsy — Enhancing percutaneous transluminal angioplasty by utilizing delivery of IVL to disrupt calcium in below the knee lesions prior to full balloon dilatation at low pressures

SUMMARY:
The RESTORE (BTK) below the knee study is a prospective, non- randomized, multi-center study for treatment of stenotic lesions with the Bolt Intravascular Lithotripsy System.

DETAILED DESCRIPTION:
The RESTORE (BTK) below the knee study is a prospective, non- randomized, multi-center study for treatment of stenotic lesions with the Bolt Intravascular Lithotripsy System that was designed to enhance percutaneous transluminal angioplasty by utilizing delivery of intravascular lithotripsy (IVL) to disrupt calcium prior to full balloon dilatation at low pressures.

ELIGIBILITY:
Key Inclusion Criteria:

* Age of subject is ≥18.
* Rutherford Clinical Category 2 - 5.
* Single or multiple target lesion(s) is/are located in a de novo artery distal to the trifurcation vessels and extends to and ends above the ankle
* Calcification is at least moderate (presence of fluoroscopic evidence of calcification: 1) on parallel sides of the vessel and 2) extending ≥ 50% the length of the lesion or absolute length ≥20mm

Exclusion Criteria:

* Target lesion is within only lower extremity vessel with < 50% stenosis.
* Significant stenosis (>50% stenosis) or occlusion of inflow tract (e.g., iliac or common femoral) not successfully treated with PTA, stent or Lithotripsy and without complications
* Planned major amputation of the target leg.
* Previously implanted stent in the treatment lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Acute reduction in percent (%) diameter stenosis of target lesion | Immediately after the intervention/procedure/surgery
  Primary Effectiveness Endpoint
Composite of new-onset Major Adverse Events (MAEs) | Within 30 days following procedure
  Primary Safety Endpoint

SECONDARY OUTCOMES:
Procedural success, defined as the ability of the Bolt IVL System to achieve a post-Lithotripsy residual diameter stenosis of ≤50% (with or without adjunctive PTA therapy or stenting) | Immediately after the intervention/procedure/surgery
  as assessed by quantitative angiography via core lab evaluation.

CONTACTS AND LOCATIONS:
Locations (4):
- Medical University of Graz, Graz, Austria
- University Hospital of Split, Split, Croatia
- Klinikum Hochsauerland GmbH, Arnsberg, Germany
- Vilnius University Hospital Santaros clinics, Vilnius, Lithuania